CLINICAL TRIAL: NCT00004914
Title: A Phase II Trial of Progressive Resistance Training (PRT) Plus Procrit for the Treatment of Anemia-Related Fatigue in Cancer Patients
Brief Title: Exercise Plus Epoetin Alfa in Treating Cancer Patients Who Have Anemia-Related Fatigue
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Supportive Care
Other Study IDs: NU 98CC7; NU-98CC7; NCI-G00-1706
Record Dates: First submitted 2000-03-07; First posted 2004-03-04 (Estimated); Last update posted 2012-06-06 (Estimated); Status verified 2012-05

CONDITIONS: Anemia; Fatigue; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; anemia; fatigue
MeSH Terms: conditions — Anemia; Fatigue | interventions — Epoetin Alfa; Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: epoetin alfa
Procedure: physical therapy

SUMMARY:
RATIONALE: Exercise may decrease anemia-related fatigue, improve strength, and build up lost muscle tissue. Epoetin alfa may help improve cancer-related anemia, energy levels, and quality of life. Exercise plus epoetin alfa may be effective treatment for anemia-related fatigue.

PURPOSE: Phase II trial to study the effectiveness of exercise plus epoetin alfa in treating cancer patients who have anemia-related fatigue.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the effect of progressive resistance training and epoetin alfa on lean body mass, fatigue, exercise tolerance, functional capacity, and total body weight in cancer patients with anemia related fatigue.

OUTLINE: Patients undergo progressive resistance training (PRT) consisting of 3 sets of 8 repetitions of concentric (lifting) and eccentric (lowering) exercises over 4-6 seconds each using bench press, arm pull, knee extension, knee flexion, and double leg press followed by 1-2 minutes of rest between sets. Patients undergo warm up and cool down periods over 10 minutes prior to and following PRT. Patients perform PRT 3 times a week for 12 weeks. Patients also receive epoetin alfa subcutaneously once weekly over 4-12 weeks in the absence of unacceptable toxicity.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study over 15 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of nonmyeloid malignancy with cancer related fatigue Anemia (hemoglobin less than 10 g/dL) No clinical or radiographic evidence of lytic bone metastases

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: ECOG 0-2 Life expectancy: Greater than 4 months Hematopoietic: See Disease Characteristics Hepatic: Not specified Renal: Not specified Other: No dementia or evidence of mental incompetence No physical handicap precluding aerobic or resistance exercise No clinical abnormality that would render exercise a risk HIV negative No contraindications to epoetin alfa Not pregnant or nursing Negative pregnancy test

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 8 weeks since prior epoetin alfa Chemotherapy: Concurrent chemotherapy allowed Endocrine therapy: Not specified Radiotherapy: Concurrent radiotherapy allowed Surgery: Not specified Other: Concurrent anticancer therapy allowed At least 1 month since prior strength training of greater than 3 hours a week

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-01; Primary Completion 2001-12 (Actual); Study Completion 2001-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie Hayden Von Roenn, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (1):
- Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois, United States